CLINICAL TRIAL: NCT00984984
Title: Randomised Double-blinded Trial Comparing Efficacy and Safety of Methylprednisolone Per os Versus IV for the Treatment of Multiple Sclerosis Relapses
Brief Title: Efficacy and Safety of Methylprednisolone Per os Versus IV for the Treatment of Multiple Sclerosis (MS) Relapses
Acronym: COPOUSEP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-000590-37; ESP/07-09
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methylprednisolone PO (Experimental)
  Interventions: Drug: methylprednisolone PO
- methylprednisolone IV (Active Comparator)
  Interventions: Drug: methylprednisolone IV

INTERVENTIONS:
Drug: methylprednisolone PO — 10 capsules Methylprednisolone 100 mg and 50 ml IV NaCl 0,9% (syringe pump 30 mn to 2 h, every day during 3 days
  Arms: methylprednisolone PO
Drug: methylprednisolone IV — IV Methylprednisolone 1 g in 50 ml NaCl 0,9% (syringe pump 30 mn to 2 h) and 10 capsules of placebo, every day during 3 days
  Arms: methylprednisolone IV

SUMMARY:
The efficacy of oral corticosteroids for the treatment of relapses of multiple sclerosis has not been proved. French neurologists treat such patients with intravenous corticosteroids. The aim of the study is to check if the efficacy of high dose oral methylprednisolone is similar to the efficacy intravenous (IV) prednisolone. The main criteria of efficacy is symptom recovery within 28 days after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 55
* informed written consent
* multiple sclerosis (Mc Donald criteria, relapsing-remitting
* EDSS before relapse : 0 to 5
* relapse : increase of 1 point or more for 1 or more functional systems of Kurtzke, with SF score most affected > 1 for all functions except for sensory (> 2); duration of symptoms > 24 h

Exclusion Criteria:

* fever
* previous relapse, and/or corticosteroid treatment < 1 month before present relapse
* first symptoms of the present relapse appeared > 15 days before inclusion
* under mitoxantrone of cyclophosphamid or natalizumab treatment
* diabetes
* infection not under control
* liver or kidney failure
* psychiatric symptoms not under control
* pregnancy
* hypersensibility to methylprednisolone

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-03; Primary Completion 2013-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
At least 1 point-reduction on Kurtzke functional scale | 28 days after beginning of corticotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Le Page, MD, Principal Investigator — Rennes University Hospital
Locations (14):
- France (14):
  - Hôpital des Armées, Brest
  - CHU Cavale Blanche, Brest
  - Centre Hospitalier de Vendée, La Roche-sur-Yon
  - Centre Hospitalier de Lannion, Lannion
  - Centre hospitalier Bretagne Sud, Lorient
  - CHU Laennec, Nantes
  - Hôpital La pitié Salpétriere, Paris
  - Centre Hospitalier de Pontivy, Pontivy
  - CH de Cornouaille, Quimper
  - Hôpital de Cornouaille, Quimper
  - Rennes University Hospital, Rennes
  - Hopital Yves Le Foll, Saint-Brieuc
  - CH Saint Malo, St-Malo
  - Centre Hospitalier Bretagne Atlantique, Vannes

REFERENCES:
- [Derived] Le Page E, Veillard D, Laplaud DA, Hamonic S, Wardi R, Lebrun C, Zagnoli F, Wiertlewski S, Deburghgraeve V, Coustans M, Edan G; COPOUSEP investigators; West Network for Excellence in Neuroscience. Oral versus intravenous high-dose methylprednisolone for treatment of relapses in patients with multiple sclerosis (COPOUSEP): a randomised, controlled, double-blind, non-inferiority trial. Lancet. 2015 Sep 5;386(9997):974-81. doi: 10.1016/S0140-6736(15)61137-0. Epub 2015 Jun 28. PMID 26135706